CLINICAL TRIAL: NCT07182604
Title: Effectiveness of a Prenatal Educational Intervention to Prevent Positional Occipital Plagiocephaly: a Randomized Multicenter Controlled Trial
Brief Title: Effectiveness of a Prenatal Educational Intervention to Prevent Positional Occipital Plagiocephaly
Acronym: POP2019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: Azienda Ospedaliero-Universitaria Careggi (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Ospedale Infermi Rimini (Unknown)
Responsible Party: Principal Investigator, Viola Fortini, Physiotherapist, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: POP2019
Record Dates: First submitted 2025-09-09; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Plagiocephaly, Positional
Keywords: plagiocephaly positional; prevention
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized intervention study with a 1:1 ratio, with cluster randomization of the dates of the monthly prenatal courses, carried out by the coordinating center for each satellite center, using a computerized system; with blinded evaluator.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Parents who received the educational program on POP prevention
  Interventions: Other: educational program on the POP prevention
- Standard of care (No Intervention): Parents who do not received the educational program on POP prevention

INTERVENTIONS:
Other: educational program on the POP prevention — During a regular prenatal class meeting, parents belonging to this group received information about POP and how to prevent it (a presentation by a physiotherapist, a video shown to all centers participating in the study, practical demonstrations of activities using a doll, and a brochure with prevention tips). The children were then assessed at birth to rule out congenital disorders and at 3 months to detect any POP and associated postural problems. They were then sent a questionnaire to assess their perceived quality of the educational intervention carried out by the physiotherapist during the prenatal course.
  Arms: Experimental group

SUMMARY:
Positional occipital plagiocephaly (POP) is a morphological abnormality of the cranium which, in the absence of early synostosis of the cranial sutures, is caused by external forces acting on the skull, which is highly malleable in newborns. The most common form of POP is the "acquired" type, which manifests around 2-3 months of age and reaches its peak severity around 4 months. The incidence of POP is 46.6% at 7-12 weeks of life, and 78.3% of cases are mild severity. In addition to being an aesthetic problem, POP can alter the first phase of a child's postural-motor development, causing postural asymmetries in the neck or spine, or asymmetries in the functional motor skills. Often, attention is only paid to the condition at a later stage, when the situation is very evident and often associated with other issues, resulting in longer, more expensive physiotherapy treatments and poorer outcomes.

Recently, interest has emerged in the possibility of preventing POP: studies have been conducted showing that preventive and educational intervention with families on the most appropriate ways of caring for their babies after birth effectively reduces the incidence and severity of POP in the first months of life and that good nationwide training of healthcare professionals on this topic could help minimize public healthcare costs.

The Specialist Interest Group (GIS) in Pediatric Physiotherapy of the AIFI Italian Association of Physiotherapists (AIFI) has produced a brochure for parents on the prevention of POP.

Primary endpoint: to assess whether the educational intervention for the prevention of POP carried out by the physiotherapist, as part of the prenatal program, reduces the incidence of POP in infants at 3 months of age.

Secondary endpoints: to assess whether the educational intervention is effective in preventing the problems often associated with POP (postural torticollis, muscle contracture in the neck, benign scoliosis, immaturity in axial control).

ELIGIBILITY:
Inclusion Criteria:

* Participation of parents in the prenatal course at 34-38 weeks of gestation;
* Signing of the informed consent form;

Exclusion Criteria:

* parents (mother or both) aged < 18 years;
* foreign parents with difficulty in understanding the Italian language and therefore giving informed consent to the study.

In addition, children who present the following conditions at birth has been excluded from the study:

* prematurity with gestational age < 36 weeks;
* neonatal distress;
* congenital occipital plagiocephaly - with cranial asymmetry measurable using a craniometer and ODDI (cranial asymmetry index) > 112.6%;
* clavicle fractures;
* congenital clubfoot, metatarsus varus;
* congenital spinal and pelvic abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Difference in the ODDI index measured with a craniometer | 0,3 months post born

SECONDARY OUTCOMES:
Difference in number of children affected by torticollis, benign scoliosis, axial immaturity in control group and intervention group | 0,3 months afther birth

CONTACTS AND LOCATIONS:
Locations (1):
- Viola Fortini, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: No